CLINICAL TRIAL: NCT00054470
Title: A Phase II Evaluation Of The Efficacy And Safety Of R115777 (NSC702818) A Non-Peptidomimetic Farnesyl Transferase Inhibitor, And Trastuzumab In Patients With Advanced Breast Cancer
Brief Title: Tipifarnib Plus Trastuzumab in Treating Patients With Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270686; U01CA069853 (NIH); P30CA054174 (NIH); SACI-IDD-01-44 (Other: San Antonio Cancer Institute); NCI-5330 (Other: NCI); UTHSC-IDD-01-44 (Other: UTHSCSA IRB)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: tipifarnib

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining tipifarnib with trastuzumab may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining tipifarnib with trastuzumab in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of tipifarnib and trastuzumab (Herceptin) in patients with metastatic breast cancer.
* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral tipifarnib twice daily on days 1-21 and trastuzumab (Herceptin) IV over 30-90 minutes on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 18-40 patients will be accrued for this study within 9-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the breast

  * HER2/neu 3+ by immunohistochemical staining

    * 2+ eligible provided HER2/neu positive by fluorescent in-situ hybridization (FISH)
    * HER2/neu positive by FISH alone allowed
* Unidimensionally measurable disease

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Must have received prior trastuzumab (Herceptin)
* Patients with known brain metastases meeting any of the following criteria are not eligible:

  * Require high-dose steroid therapy or enzyme-inducing anticonvulsant drugs
  * No prior cranial radiotherapy
  * Have progressive neurologic dysfunction that would preclude study evaluation
  * Have evidence of progressive CNS disease by CT scan or MRI
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Ejection fraction greater than 50% by MUGA or echocardiogram

Gastrointestinal

* No gastrointestinal tract disease resulting in an inability to tolerate oral medication
* No requirement for IV alimentation
* No active peptic ulcer disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant traumatic injury within the past 21 days
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No ongoing or active infection
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to tipifarnib (e.g., quinolones) or trastuzumab
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent medical illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior bone marrow transplantation with high-dose chemotherapy
* No concurrent immunotherapy

Chemotherapy

* See Biologic therapy
* No more than 2 prior chemotherapy regimens for metastatic disease
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

  * Prior combination chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* Prior hormonal therapy allowed
* No concurrent hormonal therapy for cancer

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior wide-field radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* Prior modified radical mastectomy or lumpectomy with axillary node dissection allowed
* Prior resection of metastatic lesions allowed
* More than 21 days since prior major surgery
* No prior surgery affecting absorption

Other

* No prior tipifarnib
* More than 6 weeks since initiation of bisphosphonate therapy (if bone lesions are the only site of measurable disease)
* Bisphosphonate therapy may not be initiated during study
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent antacids within 2 hours of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-12; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garry Schwartz, MD, Study Chair — Brooke Army Medical Center